CLINICAL TRIAL: NCT03490149
Title: Prediction of the Cognitive Effects of Electroconvulsive Therapy Via Machine Learning and Neuroimaging
Acronym: CoEffECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Maximilian Kiebs, M.Sc. - University Hospital Bonn (Department of Medical Psychology) (Unknown)
Responsible Party: Principal Investigator, Rene Hurlemann, Prof. Dr. Dr., University Hospital, Bonn
Other Study IDs: CoEffECT - Study
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: ECT; Depression; Cognitive Impairment; Memory Impairment
Keywords: ECT; Electroconvulsive Therapy; Depression; Memory; Memory Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ECT
  Interventions: Device: Electroconvulsive Therapy
- Medication - Treatment as usual
  Interventions: Drug: Medication - Treatment as usual
- Healthy controls

INTERVENTIONS:
Device: Electroconvulsive Therapy — Series of electroconvulsive therapy for major depressive disorder
  Groups: ECT
Drug: Medication - Treatment as usual — Medication only sample - Treatment as usual
  Groups: Medication - Treatment as usual

SUMMARY:
The study aims to use machine learning to predict the occurrence of episodic and autobiographical memory deficits as well as treatment response following a course of electroconvulsive therapy. Additionally, the neurophysiological correlates of the cognitive effects after a course of ECT will be investigated.

Therefore, structural, resting-state and diffusion tensor images will be collected within one week before the first and after the last ECT treatment from severely depressed patients. Standard measures of cognitive function and specifically episodic as well as autobiographical memory will also be collected longitudinally and used for prediction. The study consists of 60 ECT receiving inpatients suffering from major unipolar or bipolar depression, 60 medication-only controls and 60 healthy controls.

DETAILED DESCRIPTION:
Due to the immense disease burden of major depression and unsatisfactory response to standard pharmacological and psychological treatments, the need for treatment alternatives is evident. Electroconvulsive therapy (ECT) remains to be the most efficacious treatment known for treatment-resistant depression. However, although many studies show response rates above 70%, ECT can be considered vastly underused. Reasons contributing to this phenomenon may include stigma, regulatory restrictions, limited medical training, safety and side-effect concerns, or reluctance among professionals to recommend ECT. Most of these reasons have already been refuted or put into perspective by psychological and neuroscientific studies (e.g. ECT causes brain lesions) and most cognitive deficits related to the ECT course seem to fade after several weeks of discontinuation.

Still, in terms of the tolerability, memory disturbances remain the most problematic effect of ECT. Besides subjective reports from patients after a course of ECT, experimental studies have also found evidence of episodic and autobiographical memory impiarment attributable to ECT. The origins of these effects are still largely unknown and remain a goal for further research.

It has now been shown that structural T1 weighted MR-images can be used to predict the response to a course of ECT via machine learning. Therefore, this study aims to use machine learning to predict the occurrence of episodic and specifically autobiographical memory deficits arising within a course of electroconvulsive therapy based on MR-images collected within one week before the first ECT treatment from severely depressed patients. Additionally, the neurophysiological correlates of the cognitive effects modulated by a course of ECT will be investigated longitudinally through the use of structural, resting-state and diffusion tensor images. The study consists of 60 ECT receiving inpatients suffering from major unipolar or bipolar depression.

If successful, this line of research should lead to a better tolerability of ECT by aiding in the complex decision making process involved in prescribing ECT as well as the parameter setting within a treatment course (e.g. uni- vs. bilateral).

ELIGIBILITY:
Inclusion Criteria:

* The duration of the current depressive episode is at least four weeks
* The duration of the current depressive episode is less than five years
* Inpatients of the psychiatric clinic of the University Hospital Bonn and eligible for ECT because of major depressive disorder or major depressive episode in bipolar disorder (according to DSM-5 criteria)
* Score on HDRS 28 ≥ 20
* Ability to understand the purpose of and procedures required for the study and willingness to consent to participation
* Meeting of standard medical prerequisites for ECT (judged by staff psychiatrist)
* Ability to speak and understand the german language

Exclusion Criteria:

* No lifetime occurence of a personality disorder
* Current (or within the last year) posttraumatic stress disorder
* Schizophrenia or any other psychotic disorder except for psychotic depression
* Severe somatic or neurological condition (e.g. stroke)
* Head trauma resulting in unconsciousness for more than 5 minutes
* Pregnancy
* Maintenance ECT or ECT received during the last 6 month
* Subjects who do not consent to be informed of incidental findings that could have healthcare implications
* Drug or alcohol dependence (<6 month before ECT)
* Is currently enrolled in a study with an investigational study drug
* Has any condition that, in the opinion of the investigator, would compromise the wellbeing of the subject or the study or prevent the subject from meeting or performing study requirements

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients at the psychiatric hospital of the University Hospital Bonn. The patients diagnosis of major depressive disorder will be verified via the structured clinical interview for DSM-5. ECT protocol in line with international standards administered by a staff psychiatrist.
  Additionally, a medication-only and a healthy control sample are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in auditory verbal learning performance | Within one week before first and one week after last ECT
  Auditory Verbal Learning Test (AVLT)
Change in autobiographical memory performance | Within one week before first and one week after last ECT
  Autobiographical Memory Interview (AMI-SF)
Change in subjective memory impairment | Within one week before first and one week after last ECT
  Qualitative Interview
Occurence of retrograde amnesia | Within the first week after last ECT

SECONDARY OUTCOMES:
Change in depression severity as measured by the Hamilton Depression Rating Scale (HDRS 28). | One week before first and one week after last ECT
  Hamilton Depression Rating Scale (HDRS 28). Remission defined as Hamilton Depression Rating Scale-28 score of less than or equal to 9 after the ECT course. Response defined as min. -50% change in Hamilton Depression Rating Scale-28 score after ECT.
Change in depression severity as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) | One week before first and one week after last ECT
  Montgomery-Åsberg Depression Rating Scale (MADRS). Remission defined as Montgomery-Åsberg Depression Rating Scale score of less than or equal to 7 after the ECT course. Response defined as min. -50% change in Montgomery-Åsberg Depression Rating Scale score after ECT.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Hurlemann, Prof., Study Director — University Hospital, Bonn
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Sinyor M, Schaffer A, Levitt A. The sequenced treatment alternatives to relieve depression (STAR*D) trial: a review. Can J Psychiatry. 2010 Mar;55(3):126-35. doi: 10.1177/070674371005500303. PMID 20370962
- [Background] UK ECT Review Group. Efficacy and safety of electroconvulsive therapy in depressive disorders: a systematic review and meta-analysis. Lancet. 2003 Mar 8;361(9360):799-808. doi: 10.1016/S0140-6736(03)12705-5. PMID 12642045
- [Background] Haq AU, Sitzmann AF, Goldman ML, Maixner DF, Mickey BJ. Response of depression to electroconvulsive therapy: a meta-analysis of clinical predictors. J Clin Psychiatry. 2015 Oct;76(10):1374-84. doi: 10.4088/JCP.14r09528. PMID 26528644
- [Background] Sackeim HA. Modern Electroconvulsive Therapy: Vastly Improved yet Greatly Underused. JAMA Psychiatry. 2017 Aug 1;74(8):779-780. doi: 10.1001/jamapsychiatry.2017.1670. No abstract available. PMID 28658461
- [Background] Slade EP, Jahn DR, Regenold WT, Case BG. Association of Electroconvulsive Therapy With Psychiatric Readmissions in US Hospitals. JAMA Psychiatry. 2017 Aug 1;74(8):798-804. doi: 10.1001/jamapsychiatry.2017.1378. PMID 28658489
- [Background] Aoki Y, Yamaguchi S, Ando S, Sasaki N, Bernick PJ, Akiyama T. The experience of electroconvulsive therapy and its impact on associated stigma: A meta-analysis. Int J Soc Psychiatry. 2016 Dec;62(8):708-718. doi: 10.1177/0020764016675379. Epub 2016 Oct 26. PMID 27798050
- [Background] Bailine S. Reimbursement and documentation issues in an ambulatory ECT program. J ECT. 1998 Dec;14(4):255-8. PMID 9871847
- [Background] Case BG, Bertollo DN, Laska EM, Price LH, Siegel CE, Olfson M, Marcus SC. Declining use of electroconvulsive therapy in United States general hospitals. Biol Psychiatry. 2013 Jan 15;73(2):119-26. doi: 10.1016/j.biopsych.2012.09.005. Epub 2012 Oct 8. PMID 23059049
- [Background] Wilhelmy S, Rolfes V, Grozinger M, Chikere Y, Schottle S, Gross D. Knowledge and attitudes on electroconvulsive therapy in Germany: A web based survey. Psychiatry Res. 2018 Apr;262:407-412. doi: 10.1016/j.psychres.2017.09.015. Epub 2017 Sep 11. PMID 28923432
- [Background] Wilkinson D, Daoud J. The stigma and the enigma of ECT. Int J Geriatr Psychiatry. 1998 Dec;13(12):833-5. doi: 10.1002/(sici)1099-1166(1998120)13:123.0.co;2-r. No abstract available. PMID 9884906
- [Background] Dwork AJ, Arango V, Underwood M, Ilievski B, Rosoklija G, Sackeim HA, Lisanby SH. Absence of histological lesions in primate models of ECT and magnetic seizure therapy. Am J Psychiatry. 2004 Mar;161(3):576-8. doi: 10.1176/appi.ajp.161.3.576. PMID 14992989
- [Background] Semkovska M, McLoughlin DM. Objective cognitive performance associated with electroconvulsive therapy for depression: a systematic review and meta-analysis. Biol Psychiatry. 2010 Sep 15;68(6):568-77. doi: 10.1016/j.biopsych.2010.06.009. Epub 2010 Jul 31. PMID 20673880
- [Background] Payne NA, Prudic J. Electroconvulsive therapy: Part I. A perspective on the evolution and current practice of ECT. J Psychiatr Pract. 2009 Sep;15(5):346-68. doi: 10.1097/01.pra.0000361277.65468.ef. PMID 19820553
- [Background] Prudic J, Peyser S, Sackeim HA. Subjective memory complaints: a review of patient self-assessment of memory after electroconvulsive therapy. J ECT. 2000 Jun;16(2):121-32. doi: 10.1097/00124509-200006000-00004. PMID 10868322
- [Background] Lisanby SH, Maddox JH, Prudic J, Devanand DP, Sackeim HA. The effects of electroconvulsive therapy on memory of autobiographical and public events. Arch Gen Psychiatry. 2000 Jun;57(6):581-90. doi: 10.1001/archpsyc.57.6.581. PMID 10839336
- [Background] Sackeim HA. Autobiographical memory and electroconvulsive therapy: do not throw out the baby. J ECT. 2014 Sep;30(3):177-86. doi: 10.1097/YCT.0000000000000117. PMID 24755727
- [Background] Sackeim HA. Memory and ECT: from polarization to reconciliation. J ECT. 2000 Jun;16(2):87-96. doi: 10.1097/00124509-200006000-00001. No abstract available. PMID 10868319
- [Background] Redlich R, Opel N, Grotegerd D, Dohm K, Zaremba D, Burger C, Munker S, Muhlmann L, Wahl P, Heindel W, Arolt V, Alferink J, Zwanzger P, Zavorotnyy M, Kugel H, Dannlowski U. Prediction of Individual Response to Electroconvulsive Therapy via Machine Learning on Structural Magnetic Resonance Imaging Data. JAMA Psychiatry. 2016 Jun 1;73(6):557-64. doi: 10.1001/jamapsychiatry.2016.0316. PMID 27145449